CLINICAL TRIAL: NCT04049084
Title: An Observational Long-term Follow-up Study for Patients Previously Treated With Autologous ex Vivo Gene Therapy for Severe Combined Immunodeficiency Due to Adenosine Deaminase Deficiency (ADA-SCID)
Brief Title: An Observational LTFU Study for Patients Previously Treated With Autologous ex Vivo Gene Therapy for ADA-SCID
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Donald B. Kohn, M.D., Principal Investigator, University of California, Los Angeles
Other Study IDs: OTL-101-6
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Adenosine Deaminase Deficiency; Severe Combined Immunodeficiency (SCID)
Keywords: OTL-101
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Severe Combined Immunodeficiency | interventions — Genes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Biospecimen Retention: Samples With DNA — This study is a long term follow up for subjects treated with EFS ADA gene therapy via mutiple/different trials under the same IND. Samples collected from blood - cells samples, serum and DNA will be frozen and retained. Subjects followed for a period of 13 years under this Long term follow up trial post treatment and completion of the 2 year follow-up in the parent treatment trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: autologous ex vivo gene therapy products based on the EFS LV encoding for the human adenosine deaminase (ADA) gene (EFS-ADA LV) — ADA-SCID patients previously treated with autologous ex vivo gene therapy products based on the EFS LV encoding for the human adenosine deaminase (ADA) gene (EFS-ADA LV)

SUMMARY:
This observational long-term follow-up study is designed to collect safety and efficacy data from ADA-SCID patients previously treated with autologous ex vivo gene therapy products based on the EFS-ADA LV encoding for human adenosine deaminase (ADA) gene (EFS-ADA LV), as part of the OTL-101 clinical development program. No investigational medicinal product will be administered to these patients as part of the OTL-101-6 study.

DETAILED DESCRIPTION:
The overall aim of this study is to record and evaluate long-term safety and efficacy data from ADA-SCID patients previously treated with autologous ex vivo gene therapy products based on the EFS-ADA vector, as part of the UCL/A- ADA clinical development program. This will fulfil the requirements for the monitoring of delayed adverse events set by regulatory agencies for subjects treated with gene therapies.

The study will have the following specific objectives:

* To characterize the long-term safety of the gene therapy treatment;
* To characterize the long-term clinical efficacy of the gene therapy treatment. Patients who were treated as part of the UCL/A-ADA clinical development program but did not complete the expected follow- up period (e.g. as a consequence of early withdrawal due to safety events) will be included in the LTFU study, subject to their consent and compliance with inclusion and exclusion criteria.

For any patients who completed their expected follow-up period before this study became available, outcome data will be retrospectively collected for the intervening period. From the first LTFU assessment onwards, prospective data will be gathered from the annual standard of care evaluations the patients will receive from the PI or their local healthcare professionals (HCPs).

Each patient, or their legal guardian, will be required to provide informed consent, which will define the objectives of this study, the expected duration of the patient's participation, as well as the data to be collected and the schedule of collection. It is anticipated that data will be collected annually to coincide with standard of care visits.

The study outcomes will be:

* Overall survival (OS) at 15 years of follow-up post treatment with gene therapy;
* Event-free survival (EvFS) at 15 years of follow-up post treatment with gene therapy. An "event" will be defined as enzyme replacement therapy (ERT) reinstitution, need for a rescue allogeneic hematopoietic stem cell transplant (HSCT) or further gene therapy treatment;
* Use of immunoglobulin replacement therapy (IgRT);
* Adverse events (AEs), serious adverse events (SAEs) and safety concerns
* Other physical and laboratory parameters

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for enrollment in the study if all of the following criteria are met:

1. the patient has been treated with an autologous ex vivo gene therapy product based on the EFS-ADA LV, as part of the OTL-101 clinical development program;
2. the patient displays persistent detectable gene marking, as determined by the Investigator;
3. the patient or, if applicable, the patient's parent(s)/legal guardian(s), are able and willing to provide informed consent.

Exclusion Criteria:

* There are no exclusion criteria for participation in this observational LTFU study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational LTFU study is open for enrollment to ADA-SCID patients previously treated with autologous ex vivo gene therapy products based on the EFS-ADA lentiviral vector as part of the OTL-101 clinical development program. Patients treated in clinical trials as part of IND #15440, study OTL-101-5 (EudraCT No 2017-001275-23) or study 10-MI-29 (EudraCT No 2010-024253-36), as well as in Expanded Access or Compassionate Use Programs, will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2040-08 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 15 years post-treatment
  Establishing efficacy through overall survival
Event-Free Survival | 15 years post-treatment
  Establishing efficacy through event-free survival
Incidence of Adverse Events | 15 years post-treatment
  Long-Term Safety incidence of AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Donald B. Kohn, M.D., Study Director — University of Califorina, Los Angeles
Locations (2):
- Mattel Children's Hospital UCLA/Ronald Reagan UCLA Medical Center, Los Angeles, California, United States
- UCL Great Ormond Street Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth C, Masiuk K, Vazouras K, Fernandes A, Xu-Bayford J, Campo Fernandez B, Roy S, Curio-Penny B, Arnold J, Terrazas D, Reid J, Gilmour KC, Adams S, Alvarez Mediavilla E, Mhaldien L, O'Toole G, Ahmed R, Garabedian E, Malech H, De Ravin SS, Moore TB, De Oliveira S, Pellin D, Lin TY, Dang TT, Cornetta K, Hershfield MS, Hara H, Thrasher AJ, Gaspar HB, Kohn DB. Long-Term Safety and Efficacy of Gene Therapy for Adenosine Deaminase Deficiency. N Engl J Med. 2025 Oct 16;393(15):1486-1497. doi: 10.1056/NEJMoa2502754. PMID 41092330